CLINICAL TRIAL: NCT04509947
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Ad26.COV2.S in Adults
Brief Title: A Study of Ad26.COV2.S in Adults (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108871; VAC31518COV1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ad26.COV2.S: High Dose (Experimental): Participants (healthy adults aged greater than or equal to (>=) 20 to less than or equal to (<=) 55 years [cohort 1] and >= 65 years [cohort 2]) will receive intramuscular (IM) injection of Ad26.COV2.S at high dose, as 2-dose schedule on Day 1 and Day 57.
  Interventions: Biological: Ad26.COV2.S
- Ad26.COV2.S: Low Dose (Experimental): Participants (healthy adults aged >= 20 to <= 55 years [cohort 1] and >= 65 years [cohort 2]) will receive IM injection of Ad26.COV2.S at low dose, as 2-dose schedule on Day 1 and Day 57.
  Interventions: Biological: Ad26.COV2.S
- Placebo (Placebo Comparator): Participants (healthy adults aged >= 20 to <= 55 years [cohort 1] and >= 65 years [cohort 2]) will receive IM injection of placebo on Day 1 and Day 57.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.COV2.S — Ad26.COV2.S will be administered as IM injection at 2-dose (high and low) levels.
  Other Names: JNJ-78436735; Ad26COVS1
  Arms: Ad26.COV2.S: High Dose; Ad26.COV2.S: Low Dose
Biological: Placebo — Placebo will be administered as IM injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of Ad26.COV2.S administered intramuscularly (IM) at 2-dose levels, as 2-dose schedule in healthy participants aged greater than or equal to 20 to less than or equal to 55 years and greater than or equal to 65 years in good health with or without stable underlying conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI) less than (<) 40.0 kilograms per meter square (kg/m^2)
* Contraceptive (birth control) use by women should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies. Before randomization, participants who were born female must be either (a) not of childbearing potential; (b) of childbearing potential and practicing a highly effective method of contraception (failure rate of less than (<) 1 percent (%) per year when used consistently and correctly) and agrees to remain on such a method of contraception from signing the informed consent until 3 months after the last dose of study vaccine. Use of hormonal contraception should start at least 28 days before the first administration of study vaccine. The investigators should evaluate the potential for contraceptive method failure (example, noncompliance, recently initiated) in relationship to the first vaccination. Highly effective methods for this study include: (1) hormonal contraception: (i) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal); (ii) progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable); (2) intrauterine device (IUD); (3) intrauterine hormone-releasing system (IUS); (4) bilateral tubal occlusion/litigation procedure; (5) vasectomized partner (the vasectomized partner should be the sole partner for that participant; (6) sexual abstinence. Applicable to Cohort 2 only: Before randomization, a woman must be (a) postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause) or permanently sterile; and (b) not intending to conceive by any method.
* All female participants of childbearing potential must: have a negative highly sensitive urine or serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening; have a negative highly sensitive urine beta-hCG pregnancy test immediately prior to each study vaccine administration
* A male participant must agree not to donate sperm for the purpose of reproduction for a minimum 28 days after receiving the dose of study vaccine
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine

Exclusion Criteria

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigators and after consultation with the sponsor
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has a history of any neurological disorders or seizures including Guillain-Barre syndrome, with the exception of febrile seizures during childhood
* Participant previously received a coronavirus vaccine
* Participant has a positive molecular test result for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection, confirmed by polymerase chain reaction (PCR) at screening
* Participants who are at increased risk of severe coronavirus disease-2019 (COVID-19), that is, participants with moderate-to-severe asthma; chronic lung diseases such as chronic obstructive pulmonary disease (COPD) (including emphysema and chronic bronchitis), idiopathic pulmonary fibrosis and cystic fibrosis; diabetes (including type 1, type 2, or gestational); serious heart conditions, including heart failure, coronary artery disease, congenital heart disease, cardiomyopathies, and pulmonary hypertension; severe obesity; chronic kidney disease being treated with dialysis; participants who are immunocompromised (as outlined in other exclusion criteria); chronic liver disease, including cirrhosis; and participants who live in a nursing home or long-term care facility
* Participant currently working in an occupation with a high risk of exposure to SARS-CoV-2 (example, health care worker or emergency response personnel) or considered at the investigator's discretion to be at increased risk to acquire COVID-19 for any other reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local Adverse Events (AEs) for 7 days after First Vaccination | Day 8 (7 days after first vaccination on Day 1)
  Solicited local AEs are pre-defined local (at the injection site) AEs for which participants are specifically questioned and which are noted by participants in their diary for 7 days post first vaccination. Solicited local AEs are: injection site pain/tenderness, erythema, swelling and induration at the vaccination site. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product.
Number of Participants with Solicited Local AEs for 7 days after Second Vaccination | Day 64 (7 days after second vaccination on Day 57)
  Solicited local AEs are pre-defined local (at the injection site) AEs for which participants are specifically questioned and which are noted by participants in their diary for 7 days post second vaccination. Solicited local AEs are: injection site pain/tenderness, erythema, swelling and induration at the vaccination site. An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product.
Number of Participants with Solicited Systemic AEs for 7 days after First Vaccination | Day 8 (7 days after first vaccination on Day 1)
  Participants will be instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events include fatigue, headache, nausea and myalgia.
Number of Participants with Solicited Systemic AEs for 7 days after Second Vaccination | Day 64 (7 days after second vaccination on Day 57)
  Participants will be instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events include fatigue, headache, nausea and myalgia.
Number of Participants with Unsolicited AEs for 28 days after First Vaccination | Day 29 (28 days after first vaccination on Day 1)
  Number of participants with unsolicited AEs for 28 days after first vaccination will be reported. Unsolicited AEs are all AEs for which the participant is not specifically questioned.
Number of Participants with Unsolicited AEs for 28 days after Second Vaccination | Day 85 (28 days after second vaccination on Day 57)
  Number of participants with unsolicited AEs for 28 days after second vaccination will be reported. Unsolicited AEs are all AEs for which the participant is not specifically questioned.
Number of Participants with Serious Adverse Events (SAEs) | Up to 12 months
  SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.

SECONDARY OUTCOMES:
Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Neutralization as measured by Virus Neutralization Assay (VNA) | Up to 12 months
  SARS-CoV-2 neutralization will be measured by VNA to analyse the neutralizing antibodies to the wild-type virus and/or pseudovirion expressing S protein.
SARS-CoV-2-Binding Antibodies as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | Up to 12 months
  SARS-CoV-2 binding antibodies will be measured by ELISA to analyse the antibodies binding to the SARS-CoV-2 S protein.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (3):
- Japan (3):
  - Souseikai Hakata Clinic, Fukuoka
  - SOUSEIKAI PS Clinic, Fukuoka
  - Souseikai Fukuoka Mirai Hospital, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Tsuchiya Y, Tamura H, Fujii K, Numaguchi H, Toyoizumi K, Liu T, Le Gars M, Cardenas V, Eto T. Safety, reactogenicity, and immunogenicity of Ad26.COV2.S: Results of a phase 1, randomized, double-blind, placebo-controlled COVID-19 vaccine trial in Japan. Vaccine. 2023 Feb 24;41(9):1602-1610. doi: 10.1016/j.vaccine.2023.01.006. Epub 2023 Jan 5. PMID 36732164